CLINICAL TRIAL: NCT04621279
Title: COOLPRIME: Comparative Effectiveness for Cooling Prospectively Infants With Mild Encephalopathy
Brief Title: Cool Prime Comparative Effectiveness Study for Mild HIE
Acronym: COOLPRIME
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: University of California, San Francisco (Other); Children's National Research Institute (Other); Children's Hospital Los Angeles (Other); St. Louis University (Other); Stanford University (Other); University of Utah (Other); University of Pittsburgh Medical Center (Other); Children's Hospital Medical Center, Cincinnati (Other); University College Cork (Other); The Children's Hospital of San Antonio (Other); Harvard University (Other); Washington University School of Medicine (Other); Sharp HealthCare (Other); The Cleveland Clinic (Other); University of Florida Health (Other); Emory University (Other); Nationwide Children's Hospital (Other); Children's Hospital of Orange County (Other)
Responsible Party: Principal Investigator, Lina Chalak, PROFESSOR, University of Texas Southwestern Medical Center
Other Study IDs: STU-2022-0714
Record Dates: First submitted 2020-10-23; First posted 2020-11-09 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-01

CONDITIONS: Mild Hypoxic Ischemic Encephalopathy of Newborn
Keywords: mild HIE (Hypoxic Ischemic Encephalopathy); neonatal encephalopathy; brain ischemia; brain hypoxia
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Brain Ischemia; Hypoxia, Brain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mild HIE: Mild HIE identified in the first 6 hours of life according to the published PRIME study definition: newborn with evidence of encephalopathy (using the validated Sarnat Exam) NOT meeting prior cooling trials criteria.
  Interventions: Procedure: Normothermia; Procedure: Whole body therapeutic hypothermia

INTERVENTIONS:
Procedure: Normothermia — Usual care for first 72 hours for neonates with mild encephalopathy maintaining core temperature (36.5°C ± 1 C).
Procedure: Whole body therapeutic hypothermia — Whole-body therapeutic hypothermia (33.5°C ± 0.5°C) for 72 hours began by 6 hours of age for neonates with mild encephalopathy per site standard of care practice.

SUMMARY:
To determine effectiveness of therapy to improve neurodevelopmental outcomes in infants with mild HIE. To determine the adverse effects of Therapeutic Hypothermia (TH) in mild HIE on the neonate and his/her family. Determine heterogeneity of the treatment effect across key subgroups obtained in the first 6 hours after birth prior to the decision to initiate therapy.

DETAILED DESCRIPTION:
This study leverages practice variation within and across 15 participating sites to compare the effectiveness of TH versus normothermia for mild HIE on neurodevelopmental outcomes at 2 years of age.After standardizing all aspects of clinical care for mild HIE (except for TH vs. normothermia)we will enroll 460 infants with mild HIE into the longitudinal, observational comparative effectiveness study.The central aim of the comparative longitudinal cohort of mild HIE is (1) to compare the effectiveness of hypothermia to normothermia on neurodevelopmental outcomes at 2 years, (2) determine the adverse effects of TH on the infant and his/her family; and (3) determine the heterogeneity of treatment effects (moderating effect) across mild HIE subgroups as determined by physiological biomarkers obtained during the 6 hours window to initiate hypothermia. The decision to apply TH or normothermia will be entirely determined by practice parameters at each site.

ELIGIBILITY:
Inclusion Criteria:

Infants must meet all 3 inclusion criteria

1. Neonates born at ≥ 36 0/7 weeks
2. Mild Encephalopathy on neonatal neurologic exam within 6 hours after birth: defined as presence of at least 2 signs of mild, moderate, or severe encephalopathy with no more than 2 signs in the moderate or severe category.
3. Perinatal Acidosis based on at least one of the following (A or B):

   1. pH ≤ 7.00 in any cord or first infant gas (arterial, venous, or capillary) within ≤ 60 min OR base deficit ≥ 16 in any cord or first infant gas (arterial, venous or capillary) within ≤ 60 min
   2. If pH is between 7.01 and 7.15, OR base deficit is between 10 and 15.9 mmol/liter, OR blood gas is not available, an acute perinatal event is an additional criteria required (see below definition)

An acute perinatal event is defined by at least one of the following:

1. Apgar score at 10 min ≤ 5
2. Continued need for resuscitation at 10 min (chest compressions, bag mask ventilation, or positive pressure ventilation)
3. Uterine rupture, placental abruption, cord accident (prolapse, rupture, knot or tight nuchal cord)
4. maternal trauma, maternal hemorrhage, or cardiorespiratory arrest
5. fetal exsanguination from either vasa previa or feto-maternal hemorrhage, shoulder dystocia
6. Any evidence suggestive of acute perinatal event.

Infants are still eligible for enrollment in the COOLPRIME study if the cord or infant's first blood gas (arterial, venous, or capillary) is obtained >60 minutes of life.

Exclusion Criteria:

1. Gestational age at birth < 36 0/7 weeks
2. Birth weight < 1800gm
3. Head circumference <30cm
4. Congenital or chromosomal anomaly associated with abnormal neurodevelopment or death
5. Moderate or Severe HIE of 3 or more moderate or severe abnormalities on COOLPRIME Sarnat exam within 6 hours of life
6. Any seizures within first six hours of life
7. Redirection of care is being considered

Min Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Term infants ≥ 36 weeks' gestation with evidence of both perinatal event fetal acidosis and encephalopathy on exam.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of normothermia in infants as measured by Composite Bayley IV score | 22-26 months of age.
  Effectiveness of normothermia in infants is measured by Composite Bayley IV score scale, which is. an extensive formal developmental assessment tool for diagnosing developmental delays in early childhood. Possible scores range from 55- 120 where lower scores indicate worse outcome.

SECONDARY OUTCOMES:
Adverse events SAE | Discharge (approximately 7 days)
  Safety will be measured by the presence or absence of a serious adverse event (SAE) at discharge.
Parent-Infant stress and bonding as measured by MIBS | 3-4 months
  Parent-Infant stress and bonding is measured by Mother-to-infant bonding (MIBS) scale, which is a validated questionnaire with good psychometric properties that assesses the mother's feelings towards infant (bondedness) from birth to 4 months. Possible scores range from 0-3, where 0 indicates "not at all" and 3, "very much".
Parent-Infant stress and bonding as measured by IBQR | 3-4 months
  Parent-Infant stress and bonding is measured by Infant Behavior Questionnaire-Revised (IBQR) which measures differences in reactivity and regulation, and the structure of infant temperament and its relation to parental family functioning. Item scores were summed according to IBQR scoring rules to create scores on the 14 scales, with higher scores indicating greater levels of that temperament dimension.
Parent-Infant stress and bonding as measured by PSI | 3-4 months
  Parent-Infant stress and bonding is measured by Parenting Stress Index (PSI) which is an abbreviated version of the full-length test with 36 items in three domains (Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child) that combine to form a Total Stress scale, which helps identify families that are most in need of support services. In general, items are scored using the following 5-point scale: 1) SA (Strongly Agree), 2) A (Agree), 3) NS (Not Sure), 4) D (Disagree), 5) SD (Strongly Disagree). Responses to both the overall stress score and the three subscales are summed to generate representative scores, resulting the total stress score, perceptions of child behavioral problems, parenting distress, and parent-child dysfunctional interactions.

OTHER OUTCOMES:
Infant neurological integrity as measured with HNNE | Discharge
  Infant neurological integrity is measured with HNNE (Hammersmith Neonatal Neurological Exams), which is used to assess tone, spontaneous movements, reflexes, and visual and auditory attention allowing for a continuum of assessment from birth to 2 years. The maximum score for any one item is a score of 3 and the minimum is a score of 0. A subscore can be given for each section and the overall global score can be calculated by summing up all 26 items (range: 0-78), with higher scores indicating better neurological performance. The maximum global score is 78.
Infant neurological integrity as measured with HINE | 3 - 4 months
  Infant neurological integrity is measured with HINE (Hammersmith Infant Neurological Exams), which is used to assess tone, spontaneous movements, reflexes, and visual and auditory attention allowing for a continuum of assessment from birth to 2 years. The maximum score for any one item is a score of 3 and the minimum is a score of 0. A subscore can be given for each section and the overall global score can be calculated by summing up all 26 items (range: 0-78), with higher scores indicating better neurological performance. The maximum global score is 78.
Infant neurological integrity as measured with HINE | 22-26 months
  Infant neurological integrity is measured with HINE (Hammersmith Infant Neurological Exams), which is used to assess tone, spontaneous movements, reflexes, and visual and auditory attention allowing for a continuum of assessment from birth to 2 years. The maximum score for any one item is a score of 3 and the minimum is a score of 0. A subscore can be given for each section and the overall global score can be calculated by summing up all 26 items (range: 0-78), with higher scores indicating better neurological performance. The maximum global score is 78.
Behavioral tendency CBCL | 22-26 months of age.
  The Child Behavior Checklist-parent report (CBCL) will provide a profile of behavior and social functioning validated in relation to age and gender.
Composite PARCA-R | 22-26 months of age.
  The Parent Report of Children's Abilities-Revised (PARCA-R) is used against the Mental Development Index of the Bayley Scales.
IFS-R | 9-12 months
  Impact on Family Scale - Revised
IBQ-R | 9-12months
  Infant Behavior Questionnaire Revised (very short)

CONTACTS AND LOCATIONS:
Overall Officials: Lina Chalak, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Prempunpong C, Chalak LF, Garfinkle J, Shah B, Kalra V, Rollins N, Boyle R, Nguyen KA, Mir I, Pappas A, Montaldo P, Thayyil S, Sanchez PJ, Shankaran S, Laptook AR, Sant'Anna G. Prospective research on infants with mild encephalopathy: the PRIME study. J Perinatol. 2018 Jan;38(1):80-85. doi: 10.1038/jp.2017.164. Epub 2017 Nov 2. PMID 29095433
- [Background] Chalak LF, Nguyen KA, Prempunpong C, Heyne R, Thayyil S, Shankaran S, Laptook AR, Rollins N, Pappas A, Koclas L, Shah B, Montaldo P, Techasaensiri B, Sanchez PJ, Sant'Anna G. Prospective research in infants with mild encephalopathy identified in the first six hours of life: neurodevelopmental outcomes at 18-22 months. Pediatr Res. 2018 Dec;84(6):861-868. doi: 10.1038/s41390-018-0174-x. Epub 2018 Sep 13. PMID 30250303
- [Background] Chalak LF, Adams-Huet B, Sant'Anna G. A Total Sarnat Score in Mild Hypoxic-ischemic Encephalopathy Can Detect Infants at Higher Risk of Disability. J Pediatr. 2019 Nov;214:217-221.e1. doi: 10.1016/j.jpeds.2019.06.026. Epub 2019 Jul 10. PMID 31301853
- [Background] El-Dib M, Inder TE, Chalak LF, Massaro AN, Thoresen M, Gunn AJ. Should therapeutic hypothermia be offered to babies with mild neonatal encephalopathy in the first 6 h after birth? Pediatr Res. 2019 Mar;85(4):442-448. doi: 10.1038/s41390-019-0291-1. Epub 2019 Jan 16. PMID 30733613
- See also: Study website page for participants. — https://parents.coolprime.org/